CLINICAL TRIAL: NCT00870155
Title: An Open Label Follow-On Study to Assess the Ongoing Safety of MBP8298 In Subjects With Secondary Progressive Multiple Sclerosis
Brief Title: A Study for Patients With Multiple Sclerosis
Acronym: MAESTRO-02
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Negative efficacy results of the MAESTRO-01 trial
Sponsor: Eli Lilly and Company (Industry)
Collaborators: BioMS Technology Corp. (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12789; I3E-BM-MSAC; 2007-001480-30; MBP8298-SP-02
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — MBP-8298

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dirucotide (Experimental)
  Interventions: Drug: dirucotide

INTERVENTIONS:
Drug: dirucotide — 500mg, intravenous, every 6mos until regulatory approval, denial or sponsor termination
  Other Names: MBP8298; LY2820671

SUMMARY:
To obtain additional safety data in subjects who have previously completed the MBP8298-01 study "A Double Blind Placebo Controlled Multi-Centre to Evaluate the Efficacy and Safety of MBP8298 in Subjects with Secondary Multiple Sclerosis" Dirucotide is generic name for MBP8298.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects participating in this study must have completed treatment and all required evaluations in the previous MBP8298-01 study "A Double Blind Placebo Controlled Multi-Centre Study to Evaluate the Efficacy and Safety of MBP8298 in Subjects with Secondary Progressive Multiple Sclerosis",
2. Subject must be able and willing to give meaningful, written informed consent prior to participation in the trial in accordance with regulatory requirements,
3. In the Investigator's opinion, subjects must be reliable, compliant and agree to cooperate with all trial evaluations.

Exclusion Criteria:

1. Use of any concomitant disease modifying therapy for Multiple Sclerosis e.g. ß-interferon, glatiramer acetate or mitoxantrone, cyclophosphamide, methotrexate, azathioprine, or any other immuno-modulating (e.g. IVIG) or immunosuppressive drugs including recombinant or non-recombinant cytokines.
2. Any medical, psychiatric or other condition that could result in a subject not being able to give fully informed consent, or to comply with the protocol requirements.
3. Any other condition that, in the Investigator's opinion, makes the subject unsuitable for participation in the study.
4. Females who are breast feeding, pregnant or not using a medically approved method of contraception regularly.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To assess clinically significant effects of MBP8298 synthetic peptide in all subjects by collecting adverse event, ECG, laboratory, and physical exam outcomes | every 6 mos

SECONDARY OUTCOMES:
Degree of change in Kurtzke Expended Disability Status (EDSS) | every 6mos
Brain atrophy by MRI | every 6mos
Activity analysis of T2 and Gadolinium enhancing lesions | every 6mos
Lesion burden | every 6mos
Degree of change in MS Functional Composite Index (MSFC) | every 6mos
Relapse rates | every 6mos
Quality of life as measured by Short Form 36 (SF-36) or MSQoL54 | every 6mos

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9am-5pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- St. Michaels Hospital, Toronto, Ontario, Canada
- Copenhagen University Hospital, Copenhagen, Denmark
- West Tallinn Central Hospital, Tallinn, Estonia
- Terveystalo Turku Kuvantaminen, Turku, Finland
- Heinrich Heine Universitaets, Düsseldorf, North Rhine-Westphalia, Germany
- Vecmilgravis Hospital, Riga, Latvia
- Maaslandziekenhuis, Sittard, Netherlands
- Hospital Duran I Reynals, Barcelona, Spain
- Karolinska Universitetssjukhus, Stockholm, Sweden
- Walton Hospital, Liverpool, United Kingdom